CLINICAL TRIAL: NCT02671916
Title: Health and Quality of Life One Year After Discharge From the ICU: in Time Not Limited Quality Control After Intensive Medical Treatment
Brief Title: Health and Quality of Life One Year After Discharge From the Intensive Care Unit (ICU)
Acronym: QoL_ICU
Status: Terminated | Type: Observational
Why Stopped: insufficient number of replies by patients
Sponsor: Prof. Dr. med. Cristoph Haberthür (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. med. Cristoph Haberthür, Prof. Dr. med., Klinik Hirslanden, Zurich
Organization: Klinik Hirslanden, Zurich (Other)
Other Study IDs: QOL_2015_HIRS
Record Dates: First submitted 2015-08-17; First posted 2016-02-02 (Estimated); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Critically Ill
Keywords: QoL and Survival one year after ICU stay
MeSH Terms: conditions — Critical Illness | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- all patients: questionnaire for patients with ICU stay at least 5 days or longer without interruption at the ICU
  Interventions: Behavioral: questionnaire

INTERVENTIONS:
Behavioral: questionnaire — Investigation on all study patients, no Intervention, no groups

SUMMARY:
The goal is to capture the Quality of life and survival of patients one year after the stay at ICU. Data will be collected during the stay in the ICU and evaluated. One year after the ICU stay patients will be send a Quality of Life questionnaire they need to fill out and return. All data will be evaluated together.

DETAILED DESCRIPTION:
no detailled description necessary

ELIGIBILITY:
Inclusion Criteria:

* patients who are at least 5 days or longer without interruption at the ICU

Exclusion Criteria:

* patients with less than 4 days at the ICU

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all patients with conditions that lead to an ICU stay
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2015-01; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Survival | 1 year after ICU discharge

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Haberthür, MD, Principal Investigator — Klinik Hirslanden, Zurich
Locations (1):
- Klinik Hirslanden, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No